CLINICAL TRIAL: NCT01377194
Title: A Double-blind, Placebo-Controlled, Fixed-Dose Study of Levomilnacipran SR in Patients With Major Depressive Disorder
Brief Title: Safety and Efficacy of Levomilnacipran ER (Levomilnacipran SR) in Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LVM-MD-10
Record Dates: First submitted 2011-06-10; First posted 2011-06-21 (Estimated); Results first posted 2013-10-29 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-08

CONDITIONS: Major Depressive Disorder
Keywords: Depression; Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Levomilnacipran

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): 40mg Levomilnacipran ER
  Interventions: Drug: Levomilnacipran ER
- 2 (Experimental): 80mg of Levomilnacipran ER
  Interventions: Drug: Levomilnacipran ER
- 3 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levomilnacipran ER — Drug: Levomilnacipran ER 40mg/day Study drug is to be given orally, in capsule form, once daily, for 8 weeks
  Arms: 1
Drug: Levomilnacipran ER — Drug: Levomilnacipran ER 80mg/day Study drug is to be given orally, in capsule form, once daily, for 8 weeks
  Arms: 2
Drug: Placebo — Matching placebo to be given orally, in capsule form, once daily, for 8 weeks.
  Arms: 3

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and tolerability of Levomilnacipran ER compared to placebo in patients with Major Depressive Disorder (MDD).

ELIGIBILITY:
Inclusion Criteria:

* Men and women, 18-75 years old
* Currently meet the DSM-IV-TR criteria for Major Depressive Disorder
* The patient's current depressive episode must be at least 6 weeks in duration

Exclusion Criteria:

* Women who are pregnant, women who will be breastfeeding during the study, and women with childbearing potential who are not practicing a reliable method of birth control.
* Patients who are considered a suicide risk
* Patients with a history of meeting DSM-IV-TR criteria for
* a. any manic or hypomanic episode
* b. schizophrenia or any other psychotic disorder
* c. obsessive-compulsive disorder.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 568 (Actual)
Dates: Start 2011-06; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl Gommoll, MS, Study Director — Forest Research Institute, a subsidiary of Forest Laboratories
Locations (51):
- United States (47):
  - Forest Investigative Site 039, Birmingham, Alabama
  - Forest Investigative Site 037, Beverly Hills, California
  - Forest Investigative Site 012, Encino, California
  - Forest Investigative Site 038, Newport Beach, California
  - Forest Investigative Site 024, Oceanside, California
  - Forest Investigative Site 001, Redlands, California
  - Forest Investigative Site 031, San Diego, California
  - Forest Investigative Site 050, Sherman Oaks, California
  - Forest Investigative Site 034, Cromwell, Connecticut
  - Forest Investigative Site 021, Coral Springs, Florida
  - Forest Investigative Site 043, Fort Myers, Florida
  - Forest Investigative Site 018, Gainesville, Florida
  - Forest Investigative Site 060, Hallandale, Florida
  - Forest Investigative Site 020, Jacksonville, Florida
  - Forest Investigative Site 005, Ocala, Florida
  - Forest Investigative Site 014, Orlando, Florida
  - Forest Investigative Site 028, Orlando, Florida
  - Forest Investigative Site 046, Atlanta, Georgia
  - Forest Investigative Site 041, Chicago, Illinois
  - Forest Investigative Site 054, Chicago, Illinois
  - Forest Investigative Site 026, Hoffman Estates, Illinois
  - Forest Investigative Site 045, Indianapolis, Indiana
  - Forest Investigative Site 056, Prairie Village, Kansas
  - Forest Investigative Site 049, Haverhill, Massachusetts
  - Forest Investigative Site 044, Cherry Hill, New Jersey
  - Forest Investigative Site 023, Willingboro, New Jersey
  - Forest Investigative Site 004, Brooklyn, New York
  - Forest Investigative Site 002, Mount Kisco, New York
  - Forest Investigative Site 016, New York, New York
  - Forest Investigative Site 051, New York, New York
  - Forest Investigative Site 042, Orangeburg, New York
  - Forest Investigative Site 061, Raleigh, North Carolina
  - Forest Investigative Site 010, Dayton, Ohio
  - Forest Investigative Site 048, Oklahoma City, Oklahoma
  - Forest Investigative Site 053, Portland, Oregon
  - Forest Investigative Site 017, Salem, Oregon
  - Forest Investigative Site 011, Allentown, Pennsylvania
  - Forest Investigative Site 052, Bridgeville, Pennsylvania
  - Forest Investigative Site 027, Philadelphia, Pennsylvania
  - Forest Investigative Site 059, Lincoln, Rhode Island
  - Forest Investigative Site 029, Memphis, Tennessee
  - Forest Investigative Site 009, Dallas, Texas
  - Forest Investigative Site 007, San Antonio, Texas
  - Forest Investigative Site 035, San Antonio, Texas
  - Forest Investigative Site 022, Bellevue, Washington
  - Forest Investigative Site 055, Seattle, Washington
  - Forest Investigative Site 057, Spokane, Washington
- Canada (4):
  - Forest Investigative Site 025, Kelowna, British Columbia
  - Forest Investigative Site 036, Sydney, Nova Scotia
  - Forest Investigative Site 006, Chatham, Ontario
  - Forest Investigative Site 003, Ottawa, Ontario

REFERENCES:
- [Derived] Cutler AJ, Gommoll CP, Chen C, Greenberg WM, Ruth A. Levomilnacipran Extended-Release Treatment in Patients With Major Depressive Disorder: Improvements in Functional Impairment Categories. Prim Care Companion CNS Disord. 2015 Jun 11;17(3):10.4088/PCC.14m01753. doi: 10.4088/PCC.14m01753. eCollection 2015. PMID 26644957
- [Derived] Bakish D, Bose A, Gommoll C, Chen C, Nunez R, Greenberg WM, Liebowitz M, Khan A. Levomilnacipran ER 40 mg and 80 mg in patients with major depressive disorder: a phase III, randomized, double-blind, fixed-dose, placebo-controlled study. J Psychiatry Neurosci. 2014 Jan;39(1):40-9. doi: 10.1503/jpn.130040. PMID 24144196

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient recruitment occurred during a 6 month period from June to December 2011 at 47 study sites in the United States and 4 study sites in Canada.
Pre-assignment Details: All patients went through a 1-week single-blind placebo run-in period before randomization.
Groups:
- Placebo: Dose matched placebo, oral administration in capsule form, once daily for 8 weeks.
- Levomilnacipran ER 40 mg: 40mg of Levomilnacipran ER, oral administration in capsule form, once daily, for 8 weeks
- Levomilnacipran ER 80 mg: 80mg of Levomilnacipran ER, oral administration in capsule form, once daily, for 8 weeks
Period: Overall Study
Arm/Group | Placebo | Levomilnacipran ER 40 mg | Levomilnacipran ER 80 mg
Started | 186 | 188 | 188
Completed | 154 | 145 | 142
Not Completed | 32 | 43 | 46
Not completed — Adverse Event | 3 | 12 | 19
Not completed — Lack of Efficacy | 3 | 3 | 3
Not completed — Protocol Violation | 4 | 10 | 6
Not completed — Withdrawal by Subject | 8 | 10 | 7
Not completed — Lost to Follow-up | 14 | 8 | 11

BASELINE CHARACTERISTICS:
Population: The Baseline Participant population is based on the 562 randomized patients who went on to receive double-blind treatment (Safety Population).
Groups:
- Levomilnacipran ER 40 mg; Levomilnacipran 80 mg: 40mg Levomilnacipran ER, oral administration in capsule form, once daily for 8 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | Levomilnacipran ER 40 mg | Levomilnacipran 80 mg | Total
Number analyzed (Participants) | 186 | 188 | 188 | 562
Age Continuous [Mean (Standard Deviation); unit: years] | 42.3 (13.2) | 42.9 (13.4) | 43.1 (12.8) | 42.8 (13.1)
Age, Customized [Number; unit: participants]
  < 20 | 3 | 1 | 5 | 9
  ≥ 20-29 | 35 | 35 | 28 | 98
  ≥ 30-39 | 43 | 40 | 44 | 127
  ≥ 40-49 | 45 | 49 | 53 | 147
  ≥ 50-59 | 43 | 42 | 36 | 121
  ≥ 60 | 17 | 21 | 22 | 60
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116 | 117 | 124 | 357
  Male | 70 | 71 | 64 | 205
Race/Ethnicity, Customized [Number; unit: participants]
  White | 135 | 142 | 139 | 416
  Black or African-American | 35 | 37 | 36 | 108
  Asian | 7 | 4 | 3 | 14
  American Indian of Alaska Native | 3 | 0 | 0 | 3
  Native Hawaiian or other Pacific Islander | 1 | 0 | 0 | 1
  Other Race | 5 | 5 | 10 | 20
  Hispanic | 23 | 24 | 15 | 62
  Non-Hispanic | 163 | 164 | 173 | 500
Region of Enrollment [Number; unit: participants]
  United States | 177 | 183 | 180 | 540
  Canada | 9 | 5 | 8 | 22
Weight [Mean (Standard Deviation); unit: kg] | 81.60 (17.77) | 81.35 (17.09) | 81.73 (17.57) | 81.56 (17.45)
Height [Mean (Standard Deviation); unit: cm] | 168.41 (9.69) | 169.48 (9.79) | 168.63 (8.91) | 168.84 (9.47)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kilograms Per Meter Squared] | 28.67 (5.19) | 28.25 (5.17) | 28.71 (5.68) | 28.54 (5.35)

OUTCOME MEASURES:

1. Primary Outcome: Change in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score - Mixed-effects Model for Repeated Measures (MMRM) Analysis.
Description: The Montgomery-Asberg Depression Rating Scale (MADRS) rates patients on 10 items to assess feelings of sadness, lassitude, pessimism, inner tension, suicidality, reduced sleep or appetite, difficulty concentrating, and lack of interest. Each item was scored on a 7-point scale. A score of 0 indicated the absence of symptoms, and a score of 6 indicated symptoms of maximum severity. The minimum overall score possible was 0 (absence of symptoms), with a maximum overall score of 60 (maximum severity).
Time Frame: From Baseline to Week 8
Population: Of the 568 patients randomized to receive double-blind treatment, 562 patients received at least 1 dose of treatment and were included in the Safety Population, and 557 patients received at least 1 dose of treatment and had at least 1 postbaseline MADRS assessment and were included in the ITT Population.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Placebo: Dose matched placebo oral administration in capsule form, once daily, for 8 weeks.
- Levomilnacipran ER 40 mg: 40mg Levomilnacipran ER oral administration in capsule form, once daily, for 8 weeks.
- Levomilnacipran ER 80 mg: 80mg of Levomilnacipran ER oral administration in capsule form, once daily for 8 weeks
Arm/Group | Placebo | Levomilnacipran ER 40 mg | Levomilnacipran ER 80 mg
Number analyzed (Participants) | 185 | 185 | 187
Units on a scale | -11.3 (0.77) | -14.6 (0.79) | -14.4 (0.79)
Statistical Analysis 1: Comparison: Placebo vs Levomilnacipran ER 40 mg; Test type: Superiority or Other; p = 0.0027, mixed-model for repeated measures; Least squares mean difference = -3.303, 95% CI 2-sided [-5.457 to -1.148]
Statistical Analysis 2: Comparison: Placebo vs Levomilnacipran ER 80 mg; Test type: Superiority or Other; p = 0.0043, mixed-model for repeated measures; Least squares mean difference = -3.141, 95% CI 2-sided [-5.293 to -0.988]

2. Secondary Outcome: Change in Sheehan Disability Scale (SDS) Total Score
Description: The Sheehan Disability Scale (SDS) is a 3-item clinician-rated questionnaire used to evaluate impairments in the domains of work, social life/leisure, and family life/home responsibility. All items are rated on an 11-point continuum (0 = no impairment to 10 = most severe) with the total SDS score ranging from 0 (no impairment) to 30 (most severe)
Time Frame: From Baseline to Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Levomilnacipran ER 40 mg: 40mg Levomilnacipran ER, oral administration in capsule form, once daily, for 8 weeks
Arm/Group | Placebo | Levomilnacipran ER 40 mg | Levomilnacipran ER 80 mg
Number analyzed (Participants) | 185 | 185 | 187
units on a scale | -5.4 (0.66) | -7.3 (0.68) | -8.2 (0.66)
Statistical Analysis 1: Comparison: Placebo vs Levomilnacipran ER 40 mg; Test type: Superiority or Other; p = 0.0459, Mixed Models Analysis; Mixed-effects model for repeated measures; Least squares mean difference = -1.827, 95% CI 2-sided [-3.620 to -0.033]
Statistical Analysis 2: Comparison: Placebo vs Levomilnacipran ER 80 mg; Test type: Superiority or Other; p = 0.0028, Mixed Models Analysis; Mixed-effects model for repeated measures; Least squares mean difference = -2.720, 95% CI 2-sided [-4.494 to -0.946]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over a 10 month period from June 2011 to March 2012.
Description: The Serious Adverse Event data presented here is for the safety population. The Other Adverse Event data presented here is for the safety population during the 8 week double-blind treatment period.
Arm/Group | Placebo | Levomilnacipran ER 40 mg | Levomilnacipran 80 mg
Serious Adverse Events (participants affected / at risk) | 1/186 | 3/188 | 0/188
Other Adverse Events (participants affected / at risk) | 58/186 | 90/188 | 110/188
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=186) | Levomilnacipran ER 40 mg (N=188) | Levomilnacipran 80 mg (N=188)
Facial Bones Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Intussusception (Gastrointestinal disorders) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo (N=186) | Levomilnacipran ER 40 mg (N=188) | Levomilnacipran 80 mg (N=188)
Nausea (Gastrointestinal disorders) | 11 | 27 | 29
Headache (Nervous system disorders) | 16 | 22 | 25
Dry mouth (Gastrointestinal disorders) | 7 | 19 | 18
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 6 | 4 | 15
Tachycardia (Cardiac disorders) | 6 | 4 | 15
Constipation (Gastrointestinal disorders) | 4 | 13 | 12
Dizziness (Nervous system disorders) | 1 | 7 | 12
Urinary hesitation (Renal and urinary disorders) | 0 | 6 | 12
Heart rate increased (Investigations) | 0 | 13 | 11
Erectile dysfunction (Reproductive system and breast disorders) | 1/70 | 4/71 | 9/64
Upper respiratory tract infection (Infections and infestations) | 11 | 10 | 8
Diarrhoea (Gastrointestinal disorders) | 10 | 7 | 7
Testicular pain (Reproductive system and breast disorders) | 0/70 | 3/71 | 5/64

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated in this study will be the property of Forest Research Institute, Inc. An integrated clinical and statistical report will be prepared at the completion of the study.

Publication of the results by the PI will be patient to mutual agreement between the PI and Forest Research Institute, Inc.